CLINICAL TRIAL: NCT05867186
Title: Fit to Fight Childhood Cancer: an Explorative Long-term Study on Exercise and Its Influence on Physical Performance and Psychosocial Aspects in Childhood Cancer Patients During and After Cancer Treatment.
Brief Title: Fit to Fight Childhood Cancer
Acronym: Kolibri
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Joerg Faber, Univ. Prof. Dr. med. Jörg Faber, Johannes Gutenberg University Mainz
Other Study IDs: 22-02372
Record Dates: First submitted 2023-04-06; First posted 2023-05-19 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Oncology
Keywords: Paediatric exercise oncology; Precision exercise training; Childhood cancer; Quality of life; Gait; Pain; Cardiorespiratory fitness
MeSH Terms: conditions — Neoplasms; Pain | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Exercise training — Exercise training during intensive cancer treatment, maintenance therapy and aftercare. Training mainly consists of age-appropriate and personalised endurance, strength, flexibility, balance/coordination and gait training. Exercise is provided 3 to 5 times a week lasting for 45 to 60 minutes under supervision during inpatient and outpatient stays, as well as at home. At home, patients train independently according to the exercise recommendations of the exercise professionals, receive supervised telemedical exercise sessions and/or combine their training with digital tools.

SUMMARY:
The aim of the study is to investigate the influence of exercise on physical performance and psychosocial aspects in children and adolescents with cancer during and after treatment.

DETAILED DESCRIPTION:
The longitudinal, prospective and monocentric cohort study at the University Medical Centre Mainz is based on the Europe-wide, multicentre FORTEe study [NCT05289739]. The Kolibri study aims to complement the FORTEe trial. Kolibri allows the inclusion of patients who are not receiving chemotherapy and/or radiotherapy or who are undergoing oncological aftercare.

The longitudinal design of the study will allow the effects of exercise therapy on cancer-related fatigue, health-related quality of life and other psychosocial outcomes, as well as on physical function, to be monitored over the course of oncological treatment, and will provide conclusions about the effectiveness and benefits of exercise therapy. This will enable the establishment and improvement of exercise therapy protocols, as the effects of the exercise dose applied can be observed and compared over time.

The project will also validate and test the reliability of the Mainz Resilience Score in childhood cancer (MRScc) developed in the FORTEe project. The aim is to establish a validated questionnaire to assess resilience in children and adolescents with cancer, as no questionnaires are currently available.

ELIGIBILITY:
Inclusion Criteria:

* Oncological disease according to the International Classification of Childhood Cancer.
* Planned or started anti-cancer treatment (chemo- and/or radiotherapy and/or surgery) at the Clinic and Polyclinic for Paediatrics and Adolescent Medicine of the University Medical Centre of the Johannes Gutenberg University Mainz or connection to the Paediatric Oncology Centre Mainz within the framework of aftercare.
* The patient is assessed by the treating team (pediatric oncologist, exercise professional etc.) as suitable to participate in the trial, e.g. due to medical or psychological reasons.
* Existing informed consent (or assent) to participate in the study.
* The patient is not in a terminal phase of the disease.

Exclusion criteria:

* The patient is assessed by the treating team (pediatric oncologist, exercise professional etc.) as unsuitable to participate in the trial, e.g. due to medical or psychological reasons.
* After detailed information and, if necessary, having time to consider, the patient (≥ 16 years of age) did not agree to give written informed consent to participate in the trial. In the case of minor patients (<16 years of age): The legal guardians do not assume that the child/adolescent is able to freely decide on participation or to consent to participation on the basis of the information received, and do not consent to this themselves.
* The patient (and the legal guardians) has/have insufficient knowledge of the German or English language, so that it is not possible to carry out both the informed consent and interviews (in age-appropriate language).
* The patient is in a terminal phase of the disease.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible are children or adolescents from 3 to 21 years of age with a cancer diagnosis according to the International Classification of Childhood Cancer (ICCC). The term "childhood cancer" is most commonly used to designate cancer that arises in children before the age of 18 years. Since patients older than 18 years (especially in the transition phase from adolescence to young adulthood) can also have paediatric tumour entities, the upper age limit for study inclusion was set at 21 years. The Kolibri study includes patients for whom oncological treatment (regardless of the type of therapy) at the Paediatric Oncology Centre of the University Medical Centre Mainz is planned or already being carried out and who are not in the final stage of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cancer-related fatigue score at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Cancer-related fatigue measured by the Pediatric Quality of Life Inventory (PedsQL) 3.0 Multidimensional Fatigue Scale. The PedsQL Multidimensional Fatigue Scale is composed of 18 items comprising three dimensions. Scores are transformed on a scale from 0 to 100. Higher scores indicate lower fatigue.

SECONDARY OUTCOMES:
Change from baseline in the score of resilience (measured by Mainzer Resilience Scale for childhood cancer (MRScc)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Stress reactivity measured by the Mainz Resilience Score for childhood cancer (MRScc). The MRScc consists of 4 dimensions on mental health problems and 6 dimensions on stressor exposure. For both categories mental health problems and stressor exposure 4 - 400 points can be achieved. To calculate the resilience score, the category mental health problems is divided by the category stressor exposure. A score >0 means low resilience, a score < 0 means high resilience.
Change from baseline in the score of resilience (measured by the Brief Resilience Scale (BRS)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Resilience will be evaluated using the Brief Resilience Scale (BRS). BRS is a 6 item scale, the items are rated from 1 to 5. A total score is calculated by determining the sum of the individual items which result in a total score ranging from 6 to 30. A higher score means a higher resilience.
Change from baseline in the score of resilience (measured by the Child & Youth Resilience Measure-Revised (CYRM-R)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Resilience will be evaluated using the Child & Youth Resilience Measure-Revised (CYRM-R).
  The items within the measures can be directly summed to gain a total score of an individual's resilience. For the unmodified 5-point measure (with responses going from 1-5), the minimum score is 17 and the maximum score is 85. For the overall measure and subscales, higher scores indicate characteristics associated with resilience.
Change from baseline in general self-efficacy score at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  General self-efficacy will be evaluated using the General self-efficacy scale (GSE). The total score is calculated by finding the sum of the 10 items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Change from baseline in the score of physical exercise self-efficacy at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Physical self-efficacy will be evaluated using the Physical exercise self-efficacy scale (PESE). The total score is calculated by finding the sum of the 10 items. For the GSE, the total score ranges between 5 and 20, with a higher score indicating more self-efficacy.
Change from baseline in the risk status of pain-related outcomes at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Risk will be evaluated using the Pediatric Pain Screen Tool (PPST). The questionnaire consists of nine items intended to identify a patient's risk status (high, medium, or low) of poor pain-related outcome using established psychosocial prognostic factors. The PPST is adapted from the Keele STarT Back Screening Tool (SBST) and validated for the pediatric population from 8 to 18 years. The PPST contains two subscales: physical and psychosocial items. Summing all items, PPST total scores range from 0 to 9. Psychosocial subscale scores range from 0 to 5 and 0 to 4 for the physical subscale. The low risk group was defined as a PPST total score of 0 to 2 (PPST total cutoff for disability minus the PPST psychosocial subscale cutoff for psychosocial distress). For the high-risk group, a score of 3 or greater for the PPST psychosocial subscale was defined as high-risk, and last, a total PPST score greater than or equal to 3 and psychosocial subscale 0 to 2 were defined as medium risk.
Change from baseline in the subjective pain perception (measured with the face pain scale - revised (FPS-R)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  The subjective pain rating will be measured using the Face Pain Scale - Revised (FPS-R), that is a self-report measure of the actual, subjective pain intensity developed for children. The FPS-R was adapted from the Faces Pain Scale to make it possible to score the sensation of pain on the 0-to-10 metric in children and adolescents. The scale shows a close linear relationship with visual analog pain scales across the age range of 4-16 years and has already been used and validated with children and adolescents. In addition, a visual analog scale (0-10, VAS) is used to assess the current perception of pain in study participants aged 8 years and older.
Change from baseline in the subjective pain perception (measured via visual analog scale (VAS)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  In addition to the face pain scale - revised (FPS-R), a visual analog scale (0-10, VAS) is used to assess the current perception of pain in study participants aged 8 years and older.
Change from baseline in the fear of pain (parents) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Parent Fear of Pain will be measured using the Parent Fear of Pain Questionnaire (PFOPQ). The questionnaire intended to assess a parent's pain-related fears and avoidance behaviour. The total scale score reflects parents' own pain-related fear and avoidance in the context of their child's pain, and the four subscale scores reflect: Avoidance, Fear of Pain, Fear of School, and Fear of Movement. Higher scores indicate higher levels of fear. The PFOPQ will be used since Fear and avoidance have been consistently associated with poor pain-related outcomes in children.
Change from baseline in the score of pain vigilance and awareness at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Pain Vigilance and Awareness will be measured using the Pain Vigilance and Awareness Questionnaire - Child version (PVAQ-C) that consists of 14 items to assess multidimensional aspects of attention to pain sensations in children. Items are rated on a six-point scale, ranging from 0 (never) to 5 (always). Items are summed to create a total score. Attention to pain is thought to be a key mechanism influencing the experience and chronification of pain. Sustained attention to pain is thought to lead to poor outcomes in both adults and children with chronic pain.
Change from baseline in the physical activity level (measured by the Modifed Recent Physical Activity Questionnaire (mRPAQ)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Physical activity level will be evaluated using the Modifed Recent Physical Activity Questionnaire (mRPAQ).
  The duration of listed physical activities were reported (recall time: over the past 7 days). Descriptive Statistics will be performed.
Change from baseline in the physical activity level (measured by the Modified Youth Physical Activity Questionnaire (mYPAQ)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Physical activity level will be evaluated using Modified Youth Physical Activity Questionnaire (mYPAQ).
  The duration of listed physical activities were reported (recall time: over the past 7 days). Descriptive Statistics will be performed.
Change from baseline in the physical activity level (measured by the Modified Children's Physical Activity Questionnaire (mCPAQ)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Physical activity level will be evaluated using Modified Children's Physical Activity Questionnaire (mCPAQ).
  The duration of listed physical activities were reported (recall time: over the past 7 days). Descriptive Statistics will be performed.
Change from baseline in the physical activity level and behaviour (measured by half-structured interview) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  In a semi-structured interview on physical activity, qualitative data will be collected regarding activity behaviour, motivating factors and barriers to physical activity.
Change from baseline in the physical activity level and behaviour at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Current physical activity and sedentary behaviour will be objectively recorded using an accelerometer. This should be worn during the day for 7 days. Accelerometer readings with at least four valid readings (≥ 500 min/day) will be included in the analysis. The physical activity recorded by the accelerometer will be expressed in "activity counts" (counts per minute, cpm).
Change from baseline in peak oxygen uptake (VO2peak) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Cardiopulmonary Exercise Testing (CPET) will be performed during an endurance test to exhaustion to determine the peak oxygen uptake (VO2peak).
Change in functional capacity at yearly intervals from baseline up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Measured via Six Minute Walk Test (6MWT). Functional capacity is evaluated by the walked distance.
Change in submaximal endurance performance (measured by the assisted 6-minute cycling test) at yearly intervals from baseline up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Measured via assisted 6-minute cycling test (A6MCT). Endurance performance is evaluated by the cumulative revolutions after 6 minutes.
Change from baseline in motor function at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Motor function will be measured via the QUICK motor function test.
Change from baseline in lower limbs flexibility at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  A goniometer is used to measure the range of motion (ROM) during ankle flexion and extension, as well as knee and hip flexion.
Change from baseline in hamstrings flexibility at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Hamstrings flexibility will be measured via the sit and reach test.
Change from baseline in functional strength at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Functional strength will be evaluated using the sit to stand test.
Change from baseline in arm/ leg strength at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Arm and leg strength will be evaluated using a handheld dynamometer.
Change from baseline in static balance (measured by the Static Stand Test) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Static balance will be determined with the static stand test. The test requires the test person to stand on one leg for one minute. The number of contacts with the ground is counted. The static stand test has shown to be valid and reliable with children and is feasible with childhood cancer populations.
Change from baseline in functional/dynamic balance (measured by the Berg Balance Scale) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  To assess functionality in every day life the Berg Balance Scale will be used. The scale consists of 14 items that can be rated with 0 to 4 points, with 0 rating a strong impairment. A maximum of 56 points can be reached.
Change from baseline in phase angle by means of bioelectrical impedance analysis for the examination of body composition at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  A multifrequency (5, 50, 100 kHz) bioelectrical impedance analysis is performed using a phase-sensitive impedance analyser (BIAcorpus RX4004M). For this purpose, a sinusoidal alternating current with a constant intensity is applied to the patient's wrists and ankles. The phase angle (PA, ° degree) is measured by the impedance analyser as the phase shift between current and voltage. The phase angle provides conclusions about nutritional status and body composition.
Change from baseline in the score of mental health (measured by WHO (Five) Well-Being Index) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  WHO (Five) Well-Being Index (1998 version) is used to measure Mental Health.The WHO-5 consists of five statements, which respondents rate according to the scale below:
  All of the time = 5 Most of the time = 4 More than half of the time = 3 Less than half of the time = 2 Some of the time = 1 At no time = 0. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change from baseline in the score of mental health (measured by Warwick-Edinburgh Mental Well-being Scale (WEMWBS)) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is used to measure Mental Health. WEMWBS is a 14 item scale of mental well-being covering subjective well-being and psychological functioning, in which all items are worded positively and address aspects of positive mental health. The total score of the 14-item scale WEMWBS is obtained by summing the score for each of the 14 items. The scoring range for each item is from 1 - 5 and the total score is from 14-70.
Change from baseline in the score general health-related quality of life at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Health-Related Quality of Life measured by the Measurement Model for the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales questionnaire.
  On the PedsQL Generic Core Scales, for ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).
Change from baseline in the score cancer-related health-related quality of life at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  Health-Related Quality of Life measured by the Measurement Model for the Pediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module questionnaire.
  Scores are transformed to a 0 to 100 scale. Higher scores indicate lower problems.
Change from baseline in gait pattern at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  The subject's gait pattern is evaluated using a video- and sensor-based gait analysis system. The following variables will be recorded: velocity, cadence, step length, step width, single and double support and stance.
Change from baseline in functional mobility (measured by the Gillette Functional Assessment Questionnaire - Walking Scale) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  To assess patients functionality in everyday life the Gillette Functional Assessment Questionnaire - Walking Scale (FAQ) is used. The FAQ is a parent- or self-report walking scale on the patients' general ability to function in their social environment and consists of 10 items. A rating of 6 or lower indicates restricted walking abilities. A score of 10 points is considered as typical/normal.
Change from baseline in functional mobility (measured by the Functional Gait Index) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  To assess patients functionality in everyday life the Functional Gait Index (FGI) is used.
  The FGI evaluates the dynamic balance while walking. The Index consists of 10 items. Each item can be rated with a score from 0 to 3, with 0 equaling a strong impairment. No impairment in functional gait can be observed if a patient reaches the maximum of 30 points.
Change from baseline in functional mobility (measured by the Timed-up-and-go test) at yearly intervals up to 5 years | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  To assess patients functionality in everyday life the Timed-up-and-go test (TUG) will be performed.
  The TUG refers to the capacity of children and adolescents to do daily activities. The TUG measures the time in seconds required to rise from a sitting position in a standard chair, walk 3m, turn, walk back to the chair and sit down.
Information on comorbidities (including COVID-19 and its potential long-term effects) | baseline, after 1 year, after 2 years, after 3 years, after 4 years, after 5 years
  List of relevant comorbidities assessed by medical questionnaire and medical records. Descriptive Statistics will be performed.
Composite multidimensional socioeconomic status index | baseline
  Socioeconomic status will be assessed in order to perform a confounder analysis for the main outcome cancer-related fatigue.
  The calculation of the socioeconomic status index is based on the dimensions "levels of education", "occupational status" and "income". Scores for each dimension ranged from 1 to a maximum of 7. Since the 3 subscales are included in the calculation with the same weight, the socioeconomic status index can assume values between 3.0 and 21.0. Higher scores mean higher socioeconomic status.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Faber, Univ.-Prof. Dr. med., Principal Investigator — Johannes-Gutenberg-University Medical Center
Locations (1):
- Johannes-Gutenberg-University Medical Center, Mainz, Rhineland-Palatinate, Germany